CLINICAL TRIAL: NCT04457869
Title: A Phase 2, Open-label, Single-arm, Multicenter Study of F520 in Relapsed/Refractory Primary Central Nervous System Lymphoma (PCNSL) or Secondary Central Nervous System Lymphoma (SCNSL)
Brief Title: A Study of F520 in Relapsed/Refractory Primary Central Nervous System Lymphoma (PCNSL) or Secondary Central Nervous System Lymphoma (SCNSL)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shandong New Time Pharmaceutical Co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NTP-F520-003
Record Dates: First submitted 2020-07-01; First posted 2020-07-07 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-04

CONDITIONS: Primary Central Nervous System Lymphoma; Secondary Central Nervous System Lymphoma

STUDY DESIGN:
Intervention Model Description: F520
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental)
  Interventions: Drug: F520

INTERVENTIONS:
Drug: F520 — 3mg/kg every 3 weeks

SUMMARY:
It is a multi-center, prospective, open-label, two-stage optimized design, single-arm, phase II clinical study to evaluate the efficacy and safety of F520 for the treatment of Relapsed/Refractory Primary Central Nervous System Lymphoma (PCNSL) or Secondary Central Nervous System Lymphoma (SCNSL).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female of 18 Years and older;
2. Pathologically confirmed PCNSL or SCNSL of primary testicular diffuse large B-cell lymphoma (PT-DLBCL) who failed or did not respond to at least 1 line of systemic therapy; Recurrence and refractory should meet the following definitions:

   * PCNSL patients: relapse is defined as the appearance of new lesions at the primary site or other sites after the standard treatment with MTX reaches complete remission (CR). Refractory patients were defined as those who did not reach PR in 2 cycles or CR in 4 cycles after standard treatment with MTX. If the best effect or end cause was PD, the number of courses was not required;
   * patients with SCNSL: Patients with relapsed/refractory primary testicular diffuse large B-cell lymphoma who must include central nervous system invasion. Relapse was defined as the patients who had been prevented or treated with MTX; refractory was defined as the patients who had received the latest chemotherapy regimen for 2 cycles without PR or 4 cycles without CR. if the best effect or end cause was PD, the number of courses was not required;
3. Measurable disease requirements on scans: subjects should have at least one measurable extranodal brain lesion more than 10×10mm;
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0~2;
5. Agree to provide archived tumor tissue specimens or fresh tissue specimens;
6. Life expectancy ≥ 3 months;
7. Adequate laboratory parameters during the screening period as evidenced by the following（No blood components and cell growth factors are allowed within 14 days prior to screening）:

   routine blood tests: Absolute neutrophil count ≥1.5×109/L ;Platelets ≥100×109/L;Hemoglobin ≥ 9.0 g/dL; Liver function：Total bilirubin (TBIL) ≤1.5×upper limit of normal (ULN), ALT and AST ≤2.5ULN; for subjects with liver metastases, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 5×ULN, Total bilirubin (TBIL) ≤3×upper limit of normal (ULN); Renal function CCr≤1.5×ULN，Creatinine clearance≥50 mL/min; Thyroid function indicators: thyroid-stimulating hormone (TSH) and free thyroxine (FT3/FT4) are within the normal range or no clinical significant;
8. International Normalized Ratio (INR) ≤ 1.5 and PTT (aPTT) ≤ 1.5 times the upper limit of normal;
9. Understand study procedures and contents, and voluntarily sign the written informed consent form.

Exclusion Criteria:

1. a）Patients with suspected or existing eye tumors; b）patients who cannot undergo MRI assessments c) PCNSL patients with systemic disease;
2. Patients with certain diseases such as active autoimmune disease, type I diabetes, hypothyroidism that needs hormone replacement, active infection, psychiatric disorder (Except for mild cognitive impairment caused by tumor);
3. Prior malignancy active within the previous 3 years except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast;
4. Patients with stroke within 6 months before the first dose (except for those with "multiple lacunar infarction" indicated by imaging examination, but no need for treatment) or with a history of intracranial hemorrhage (except for intracranial hemorrhage after surgery);
5. Prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways;
6. Concurrent medical condition requiring the use of immunosuppressive medications, or immunosuppressive doses of systemic or absorbable topical corticosteroids. Doses > 10 mg/day prednisone or equivalent are prohibited within 14 days before the first dose;
7. Active infection（needing therapy） or an unexplained fever > 38.5°C during screening or before the first scheduled day of dosing (subjects with tumor fever may be enrolled at the discretion of the investigator);
8. Those who received systemic therapy of radiotherapy, chemotherapy, hormone therapy, surgery, targeted therapy, or antibody drugs within 4 weeks before the first dose; used monoclonal antibody coupled radionuclide or cytotoxic therapy within 10 weeks before the first dose; the toxicity of previous anti-tumor therapy has not recovered to ≤1 (except hair loss);
9. Patients who have a history of organ transplantation or allogeneic bone marrow transplantation or who have received auto stem cell transplantation or other severe immune defects within 3 months before the first dose;
10. Patients who are preparing for autologous stem cell transplantation.
11. Patients with active pulmonary tuberculosis;
12. Previous or simultaneous interstitial lung disease (except for interstitial lung disease caused by radiotherapy and chemotherapy and without symptoms at present);
13. Patients with active hepatitis;
14. Patients with HIV positive;
15. Patients received any other clinical trial drug / device treatment within 4 weeks before the first administration;
16. Patients with uncontrollable or serious cardiovascular diseases, cardiovascular diseases such as congestive heart failure, unstable angina pectoris, myocardial infarction and other cardiovascular diseases of NYHA grade II or above occurred within 6 months before the first dose; uncontrolled hypertension (systolic pressure ≥ 180mmhg and / or diastolic pressure ≥ 100mmhg);
17. Patients with drug abuse history or alcohol addiction history within 6 months before the study drug administration;
18. Patients with known previous allergies to macromolecular protein preparations or known to be allergic to anti-PD-1 / PD-L1 antibodies
19. Patients who received live attenuated vaccine within 4 weeks before the first dose (except inactivated influenza vaccine such as seasonal influenza vaccine for injection);
20. Female and male who have reproductive potential must be willing and able to employ a highly effective method of birth control/contraception to prevent pregnancy while on treatment and for at least 6 months after receiving the last dose of study treatment.
21. The investigators judged that it was not suitable for the patients to participating in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2022-07-31 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) by Independent Review Committee (IRC) Independent Review Committee (IRC). | Approximately 24 months
  Response assessment will be performed according to modified IPCG response. criteria on contrastenhanced cranial MRI-scans.

SECONDARY OUTCOMES:
Objective response rate (ORR) based on the investigator assessment. | Approximately 24 months
  Response assessment will be performed according to modified IPCG response.
Progression-free survival (PFS) | Approximately 24 months
  Based on IRC and the investigator assessments.
Duration of response (DOR) | Approximately 24 months
  Based on IRC and the investigator assessments.
Overall survival (OS) | Approximately 24 months
Safety of F520 | Approximately 24 months
  AE/SAE will be assessed by CTCAE v5.0